CLINICAL TRIAL: NCT04993456
Title: Division of Cardiology, Department of Internal Medicne, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan 430030, China
Brief Title: Calcitonin Level and New-onset of Post-Operative Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Li Ni, Division of Cardiology, Department of Internal Medicne, Tongji Hospital
Other Study IDs: TJ-CT-POAF
Record Dates: First submitted 2021-06-24; First posted 2021-08-06 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Calcitonin Secretion Disorder; Post-operative Atrial Fibrillation
Keywords: Post-operative atrial fibrillation; Calcitonin; Cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAF group: the patients will have atrial fibrillation following the cardiac surgery
  Interventions: Procedure: Caridac surgery
- non-POAF group: the patients will have no atrial fibrillation following the cardiac surgery
  Interventions: Procedure: Caridac surgery

INTERVENTIONS:
Procedure: Caridac surgery — Cardiac surgery

SUMMARY:
Post-operative atrial fibrillation (POAF) is one of the common complicaiton following cardiac surgery, occurring in approximately 20%-40% patients. Although POAF is associated with longer hospital stays, most POAF is short lived and resolves in the 2-4 days afer cardiac surgery.

However, a recent meta-analysis showed significant increases in 1,5, and 10 year mortality in POAF patients (odds ratio:1.60, 2.60, 1.51;95% confidence intervals: 1.52 to 1.68, 2.00 to 3.38, 1.43 to 1.60;P <0.0001), the combined adjusted risk of death (16 studies, n =84,295) was also significantly increased in patients with POAF (hazard ratio: 1.25;95% confidence interval: 1.2-1.3;P < 0.0001).

These data highlight the need to understand better the underlying mechanism of POAF. A latest research in Nature reported levels of circulating calcitonin (CT), which is the main risk factor for atrial fibrillation (AF). Global disruption of CT receptor signalling in mice causes atrial fibrosis and increases susceptibility to AF.

Here we will explore the relationship between CT and POAF.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of no history of atrial fibrillation/flutter;
* 2. Heart rate ≥50 beats/min;
* 3. EF > 40%;
* 4. No history of emergency cardiac surgery in our hospital;
* 5. Participate voluntarily and sign the informed consent, and can accept the follow-up of more than 2 years.

Exclusion Criteria:

* 1. Atrial fibrillation/flutter;
* 2. Left atrial diameter >5.5cm;
* 3. Previous cardiac surgery or emergency surgery (<12h);
* 4. Sick sinus node syndrome;
* 5. Ventricular preexcitation or preexcitation syndrome;
* 6. Second degree or above atrioventricular block;
* 7.Myocardial infarction occurred within 7 days;
* 8. Infection, sepsis, rheumatic or inflammatory diseases;
* 9. Abnormal liver and kidney function (three times higher than the upper limit of normal);
* 10. Uncontrolled hyperthyroidism, severe obstructive sleep apnea, and acute alcoholism;
* 11. Any ischemic events (stroke or TIA) that occurred 180 days before the participant signed the informed consent, or any known unresolved complications from previous stroke/TIA;Thrombosis;
* 12. Patients with other diseases requiring radiotherapy, chemotherapy and long-term hormone therapy;
* 13. Patients' life expectancy makes it unlikely that follow-up will be completed;
* 14. Participate in, or are expected to participate in, other clinical trials of any drugs, devices or biologics during the study period;
* 15. Patients with contraindications to dynamic electrocardiogram;
* 16. Patients who are unwilling or unable to fully comply with study procedures and follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected that 200 patients who received the first non-emergency cardiopulmonary bypass cardiac surgery in our hospital will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
POAF lasting longer than 30 seconds during the first week after cardiac surgery | 2 years after cardiac surgery
  The incidence of atrial fibrillation lasting longer than 30 seconds during the first week after cardiac surgery

SECONDARY OUTCOMES:
The hospitalization days | 2 years after cardiac surgery
  The length of stay after the cardiac surgery
Ventricular rate of the atrial fibrillation | 2 years after cardiac surgery
  Ventricular rate of atrial fibrillation after the cardiac surgery
Levels of serum calcitonin | 2 years after cardiac surgery
  Levels of serum calcitonin of atrial fibrillation after the cardiac surgery
Levels of serum procalcitonin | 2 years after cardiac surgery
  Levels of serum procalcitonin of atrial fibrillation after the cardiac surgery
Levels of serum hsCRP | 2 years after cardiac surgery
  Levels of serum hsCRP of atrial fibrillation after the cardiac surgery
Levels of serum cytokines(IL-1β，IL-2R，IL-6，IL-8，IL-10，TNF-α) | 2 years after cardiac surgery
  Levels of serum cytokines(IL-1β，IL-2R，IL-6，IL-8，IL-10，TNF-α) of atrial fibrillation after the cardiac surgery
Atrial fibrillation burden after cardiac surgery | lidan2014@tjh.tjmu.edu.cn
  Time and length of atrial fibrillation after cardiac surgery

OTHER OUTCOMES:
Thromboembolic stroke | 2 years after cardiac surgery
  Thromboembolic stroke
Serious bleeding events | 2 years after cardiac surgery
  Serious bleeding events
All-cause mortality | 2 years after cardiac surgery
  Cardiovascular, noncardiovascular or undetermined cause of death
Recurrence atrial fibrillaiton and readmission | 2 years after cardiac surgery
  Recurrence atrial fibrillaiton and readmission

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided